CLINICAL TRIAL: NCT00439569
Title: Phase I/IIa Clinical Trial of Sodium Phenylbutyrate in Pediatric Subjects With Type II/III Spinal Muscular Atrophy
Brief Title: Clinical Trial of Sodium Phenylbutyrate in Children With Spinal Muscular Atrophy Types II or III
Acronym: NPTUNE01
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to poor compliance with study drug administration.
Sponsor: Westat (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: René Gonin, PhD (Math. Stats.), Senior Biostatistician and NPTUNE Principal Investigator, Westat
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01NS42361_NPTUNE01; HHSN265200423611C (Other Grant/Funding Number: NIH Contract); N01NS42361 (NIH)
Record Dates: First submitted 2007-02-21; First posted 2007-02-23 (Estimated); Results first posted 2010-02-12 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2009-08

CONDITIONS: Spinal Muscular Atrophy Type II; Spinal Muscular Atrophy Type III
Keywords: spinal muscular atrophy type II/III; SMA type II/III; spinal muscular atrophy; SMA; sodium phenylbutyrate; motor neuron disease; neuromuscular; survival motor neuron; SMN; dose escalation
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Muscular Atrophy, Spinal; Motor Neuron Disease | interventions — 4-phenylbutyric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Cohorts of 3 subjects were to be enrolled sequentially in escalating dosage levels. The first three subjects enrolled at 500 mg/kg/day for the duration of the study drug period. The dosage of the next cohort was determined by the Modified Continual Re-assessment Method (MCRM) calculation and approval of the Study Monitoring Committee (SMC). The MCRM calculation could indicate that additional subjects should be enrolled at the same dosage or a higher dosage.
  Interventions: Drug: sodium phenylbutyrate

INTERVENTIONS:
Drug: sodium phenylbutyrate — 500 mg/kg/day, depending upon tolerability subsequent dosages may increase to 675, 900, or 1200 mg/kg/day to identify maximum tolerated dose (MTD) and then an additional 6 participants will enroll at the MTD

SUMMARY:
The purpose of this study is to identify the maximum tolerated dosage of sodium phenylbutyrate in children with spinal muscular atrophy types II or III; and to determine if the drug has an effect on SMN mRNA and protein levels.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is a genetic, neuromuscular disorder caused by progressive degeneration of motor neurons in the spinal cord, which results from the loss of survival motor neuron (SMN) protein. The disorder is characterized by weakness and wasting of the voluntary muscles and is a leading cause of hereditary infant death. Sodium phenylbutyrate--a drug used to treat urea cycle disorders--may increase the amount of SMN protein in the body and consequently may decrease the severity of SMA. However, this has not yet been proven.

In this multicenter trial, physicians will evaluate multiple dosage levels of sodium phenylbutyrate to determine the maximum tolerated dose (MTD), or the highest dose that can be safely given to children with SMA types II or III. The initial dosage tested will be 500 mg/kg/day. Depending upon tolerability, subsequent groups may receive dosages of 675, 900, or 1200 mg/kg/day. Blood levels of SMN mRNA and protein will also be measured to determine whether sodium phenylbutyrate can increase the amount of these two biomarkers in the blood. Up to 24 children will be enrolled in the study and will be on sodium phenylbutyrate for 12 weeks. The MTD will be determined based on safety data from Day 0 through the Day 29 visit. Participants will continue to be monitored for safety and SMN mRNA and protein levels through the 12 week study drug administration period.

Potential participants will be screened by having their complete medical and treatment histories recorded, as well as undergoing a physical examination, laboratory tests, and an electrocardiogram (EKG). Parents of eligible participants will receive a supply of sodium phenylbutyrate and instructions on how to administer the drug. Participants will return to the clinic on days 8, 22, 29, and at weeks 8 and 12 of the study to update their medical and treatment histories, have a physical exam, and have blood and urine collected for laboratory testing. A follow-up clinic visit will occur approximately 14 days after the last dose of sodium phenylbutyrate is given. During this visit participants will update their complete medical and treatment histories and have a physical examination. Duration of the study is about 14 weeks.

Information from this study, which is part of the NINDS Pilot Therapeutics Network (NPTUNE), may be used for future studies to determine if sodium phenylbutyrate is effective for treating SMA, and if the drug has an effect on SMA symptoms.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria within 14 days prior to receiving the first dose of study drug.

* Weakness and hypotonia consistent with a clinical diagnosis of spinal muscular atrophy (SMA) type II or III
* Laboratory documentation of homozygous absence of SMN1 exon 7
* Type III subjects who are unable to get up from the floor unaided. "Unaided" is defined as not using a device or obtaining assistance from another person.
* 2 years of age or older, but younger than 12 years of age, at the time of enrollment
* Written informed consent of parents/guardian
* Weight greater than or equal to 10 kilograms
* Laboratory results drawn within 14 days prior to start of study drug demonstrating: Hemoglobin within normal range at the clinical site; White Blood Cell Count ≥ 3000/mm³; Platelet Count ≥ 75,000/mm³; Lipase and Amylase ≤ 1.5 x upper limit of normal (ULN) in the absence of associated clinical symptoms; AST and ALT ≤ 2.5 x ULN; Bilirubin ≤ 1.5x ULN in the absence of associated clinical symptoms; Sodium ≥ 130 and ≤ 150 mmol/L; Potassium ≥3.0 and ≤ 5.5 mmol/L; Chloride ≤ 110 mmol/L; Calcium ≥ 8.0 mg/dL; Bicarbonate ≥ 16 mmol/L; Glucose ≥ 55 and ≤ 160 mg/dL; BUN ≤ 39 mg/dL; Creatinine ≤ 1.5 x ULN
* Subject is expected to survive for at least 6 months following study entry.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participating in the study:

* Evidence of renal dysfunction, blood dyscrasia, hepatic insufficiency, symptomatic pancreatitis, cardiac arrhythmia, congenital heart defect, known history of metabolic acidosis, hypertension, significant central nervous system impairment, or neurodegenerative or neuromuscular disease other than SMA.
* Any adverse event ≥ Grade 3 at the time of screening based on the protocol toxicity grading table
* Any acute co-morbid condition interfering with the well-being of the subject within 7 days of enrollment including bacterial infection, viral infectious process, food poisoning, temperature > 99.0ºF, need for acute treatment or observation due to any other reason, as judged by the investigator
* ≥ Grade 2 vomiting;
* ≥ Grade 2 liver dysfunction/failure (clinical);
* Any abnormality noted on EKG except for asymptomatic sinus arrhythmia
* History of allergy/sensitivity to sodium phenylbutyrate
* Use of sodium phenylbutyrate within 30 days of study entry
* Serious illness requiring systemic treatment and/or hospitalization within 14 days prior to study entry (Subjects are not eligible following serious illness until therapy is complete and the subject is stable, or until the subject is on therapy and stable for at least 14 days.)
* Use of medications intended for the treatment of SMA including riluzole, valproic acid, hydroxyurea, oral use of albuterol, sodium phenylbutyrate, butyrate derivatives, creatine, carnitine, growth hormone, anabolic steroids, probenecid, oral or parenteral use of corticosteroids at entry, haloperidol, agents anticipated to increase or decrease muscle strength or agents with known or presumed histone deacetylase (HDAC) inhibition within 30 days prior to study entry

Notes: Subjects who use a nebulizer or require an inhaler to receive albuterol will be allowed in the study; however oral use of albuterol is prohibited. Topical use of steroids will be allowed. Oral use of steroids is not allowed at entry, but these may be used as clinically indicated while on study. Event grading will be based on the toxicity-grading table in the protocol.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: René Gonin, PhD, Principal Investigator — Mathematical Statistician, Westat; Peter R. Gilbert, ScM, Study Director — National Institute of Neurological Disorders and Stroke, Program Director
Locations (5):
- United States (5):
  - Stanford University Medical Center, 300 Pasteur Drive, Room A343, Stanford, California
  - Washington University Medical School, Washington University, 660 S. Euclid Avenue, Box 8111, St Louis, Missouri
  - Columbia University, 180 Fort Washington Avenue, 5th Floor, New York, New York
  - The Children's Hospital of Philadelphia, Clinical Trials Office, A-230, 34th St. and Civic Center Boulevard, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center at Dallas, Division of Pediatric Neurology, Children's Medical Center of Dallas, Ambulatory Care Pavilion, 2350 Stemmons Freeway, Suite #5074, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol was open for recruitment between January 31, 2007 and September 23, 2008 at neurology clinics affiliated with university hospitals.
Pre-assignment Details: Pre-specified dosage levels of sodium phenylbutyrate (NaPB) were calculated using the modified Fibonacci rule yielding dosage levels of 500, 675, 900 and 1200 mg /kg/day. The selection of 500 mg/kg/day as the initial dosage was based on the recommended dosage of 450 -600 mg/kg/day for the approved indication for urea cycle disorders in children.
Groups:
- Subjects Enrolled: Cohorts of 3 subjects were to be enrolled sequentially in escalating dosage levels. The first 3 subjects enrolled at 500 mg/kg/day for the duration of the study drug period. The next cohort's dosage was determined by the Modified Continual Re-assessment Method (MCRM)approach and approval of the Study Monitoring Committee (SMC). The MCRM calculation could indicate that additional subjects should be enrolled at the same dosage or a higher dosage. Due to the replacement of subjects (4 not completed), more than 3 subjects were enrolled in Cohort 1. Two new subjects were then enrolled in Cohort 2.
Period: Cohort 1 (500 mg/kg/Day)
Arm/Group | Subjects Enrolled
Started | 7
Completed | 3
Not Completed | 4
Not completed — Allergic reaction | 1
Not completed — Less than 80% study drug compliance | 3
Period: Cohort 2 (500 mg/kg/Day)
Arm/Group | Subjects Enrolled
Started | 2 (2 new subjects in Cohort 2 were enrolled into the study after Cohort 1 completed the study.)
Completed | 1
Not Completed | 1
Not completed — Less than 80% study drug compliance | 1

BASELINE CHARACTERISTICS:
Groups:
- Subjects Enrolled (Cohort 1, Cohort 2): Cohorts of 3 subjects were to be enrolled sequentially in escalating dosage levels. The first 3 subjects enrolled at 500 mg/kg/day for the duration of the study drug period. The next cohort's dosage was determined by the Modified Continual Re-assessment Method (MCRM)approach and approval of the Study Monitoring Committee (SMC). The MCRM calculation could indicate that additional subjects should be enrolled at the same dosage or a higher dosage. Due to the replacement of subjects (4 not completed), more than 3 subjects were enrolled in Cohort 1.
Arm/Group | Subjects Enrolled (Cohort 1, Cohort 2)
Number analyzed (Participants) | 9
Age, Customized [Number; unit: Participants]
  24 - 48 months | 5
  49 -96 months | 3
  >96 and < 144 months | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities (DLT)
Description: Number of DLTs to determine the maximum tolerated dosage. A DLT is defined as any Grade (GR)3 or higher adverse event(AE),GR 1 or higher cardiac arrhythmia;GR 2 or higher vomiting;GR 2 or higher liver dysfunction/failure (clinical);GR 2 elevation of amylase or lipase accompanied by clinical symptoms of pancreatitis.The following GR 2 events are classified as DLTs if evaluated to be clinically significant by the principal investigator or medical safety monitor:decrease of hemoglobin, WBCs, platelets; elevation of AST, ALT,bilirubin;abnormality of Na, K, Cl, Ca, HCO3, glucose, BUN or creatinine.
Time Frame: 29 Days
Population: The study was closed prematurely due to poor compliance with study drug administration. The MTD could not be determined as it was less than the lowest dosage studied (500 mg/kg/day).
Measure: Number; unit: DLT(s)
Arm/Group | Subjects Enrolled (Cohort 1, Cohort 2)
Number analyzed (Participants) | 0

2. Primary Outcome: Survival Motor Neuron (SMN) Messenger Ribonucleic Acid (mRNA)
Description: The change of level in blood SMN mRNA from baseline to assess time course and dose response.
Time Frame: Baseline - 12 weeks
Population: The study was closed prematurely due to poor compliance with study drug administration. These data have not yet been analyzed. Their interpretability will be limited because of the small number of specimens collected.
Measure: Mean (Standard Error); unit: Change in mRNA level
Arm/Group | Subjects Enrolled (Cohort 1, Cohort 2)
Number analyzed (Participants) | 0

3. Secondary Outcome: Drug Safety
Description: Adverse event(AE)monitoring
Time Frame: 14 weeks
Population: The study was closed prematurely due to poor compliance with study drug administration. These data have not yet been analyzed. Their interpretability will be limited because of the small number of subjects enrolled. There were no safety concerns reported by the study monitoring committee (SMC).
Measure: Number; unit: Adverse Events
Arm/Group | Subjects Enrolled (Cohort 1, Cohort 2)
Number analyzed (Participants) | 0

4. Secondary Outcome: Pharmacokinetic Parameters (Maximum Plasma Concentration)
Description: Maximum Plasma Concentration (Cmax)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Subjects Enrolled (Cohort 1, Cohort 2)
Number analyzed (Participants) | 0

5. Secondary Outcome: Pharmacokinetic Parameters (Time to Maximum Concentration)
Description: Time to Maximum Concentration (Tmax)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Subjects Enrolled (Cohort 1, Cohort 2)
Number analyzed (Participants) | 0

6. Primary Outcome: Survival Motor Neuron (SMN) Protein
Description: The change of level in blood SMN protein from baseline to assess time course and dose response.
Time Frame: Baseline - 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in SMN Protein level
Arm/Group | Subjects Enrolled (Cohort 1, Cohort 2)
Number analyzed (Participants) | 0

7. Secondary Outcome: Pharmacokinetic Parameters (Area Under the Plasma Concentration Versus Time Curve (AUC))
Description: Area Under the Plasma Concentration versus Time curve (AUC)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: µmol/L * hours
Arm/Group | Subjects Enrolled (Cohort 1, Cohort 2)
Number analyzed (Participants) | 0

8. Secondary Outcome: Overall Study Drug Compliance
Description: Subjects receiving 80% or more of the prescribed doses within each study visit interval were considered compliant.
Time Frame: 12 Weeks
Population: Four of the nine subjects enrolled were less than 80% compliant. The study was closed prematurely due to poor compliance with study drug administration.
Measure: Number; unit: Participants
Arm/Group | Subjects Enrolled (Cohort 1, Cohort 2)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Data were collected over a 17 month period
Description: Data were collected at scheduled clinic and telephone study visits via medical history, physical examinations, laboratory tests, EKG, and other tests as necessary. In addition, adverse events were reported to site investigators by subjects' parents in between visits, as needed.
Groups:
- Cohorts 1 & 2 (500 mg/kg/Day): Cohort 1 was assigned a dosage of 500 mg/kg/day. One subject was replaced due to an allergic reaction and four subjects due to less than 80 percent study drug compliance. Due to these replacements, more than 3 subjects were enrolled in the first cohort. Cohort 2 was assigned a dosage of 500 mg/kg/day by the MCRM and approved by the SMC due to dose-limiting toxicities experienced in Cohort 1. For the purpose of reporting adverse events, these two cohorts were combined for a total of 9 enrolled subjects.
Arm/Group | Cohorts 1 & 2 (500 mg/kg/Day)
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohorts 1 & 2 (500 mg/kg/Day) (N=9)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohorts 1 & 2 (500 mg/kg/Day) (N=9)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Blood bicarbonate decreased (Investigations) | 2 (2)
Blood chloride increased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 2 (2)
Chapped lips (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 1 (3)
Fatigue (General disorders) | 2 (4)
Flatulence (Gastrointestinal disorders) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2)
Increased appetite (Metabolism and nutrition disorders) | 1 (1)
Infantile spitting up (Gastrointestinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3)
Otitis media (Infections and infestations) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
The study was closed early due to poor study drug compliance. The sample size is therefore extremely limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Publication Policy for the National Institute of Neurological Disorders and Stroke (NINDS) Pilot Therapeutic Trials Network (NPTUNE) outlines procedures for the development and review of concept sheets, abstracts, publications,presentations. Investigators must submit an application to the NPTUNE Publications Committee for the use of data. A Writing Committee, appointed by the Publications Committee,is responsible for initiating, coordinating, and approving publications and presentations.